CLINICAL TRIAL: NCT06150183
Title: A First-in-Human, Open-label, Dose Escalation Trial With Expansion Cohorts to Evaluate the Safety and Preliminary Efficacy of BNT314 as Monotherapy in Patients With Advanced Malignant Solid Tumors
Brief Title: Safety and Preliminary Efficacy of BNT314 in Cancer Patients With Malignant Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT314-01; 2023-506053-38-00 (EU CTIS Number); 1008686 (Other: Integrated Research Application System (UK))
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Tumor
Keywords: Malignant solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BNT314 Monotherapy (Experimental): Escalating dose levels and backfill cohorts
  Interventions: Biological: BNT314

INTERVENTIONS:
Biological: BNT314 — Intravenous infusion

SUMMARY:
The purpose of this first-in-human study is to find out if BNT314 is safe when it is used alone in patients with different types of cancer.

This is a dose escalation study in which patients will be assigned to multiple dose levels (DLs) of BNT314 given alone. By escalating the dose with a small group of patients, the Maximum Tolerated Dose which is the highest dose with acceptable safety and manageable side effects, or the maximum administered dose will be investigated.

DETAILED DESCRIPTION:
This is a multicenter, multinational safety study in patients with metastatic or advanced malignant solid tumors for whom, at the discretion of the investigator, there is no available standard therapy likely to confer clinical benefit, evaluating the safety, tolerability, preliminary antitumor activity, pharmacokinetics (PK), pharmacodynamics, and immunogenicity of BNT314.

During dose escalation, BNT314 will be administered to patients via one infusion in periodic cycles.

Additional cohorts (backfill cohorts) administering BNT314 as monotherapy will assign patients to specific DLs, based on the emerging safety, PK, and pharmacodynamic data. This would allow for further assessment of dose- and exposure-response relationships for clinical activity, safety, and tolerability to support BNT314 dose optimization.

The treatment period will last until progressive disease (PD), confirmed PD (as per immune Response Evaluation Criteria in Solid Tumors [iRECIST]), unacceptable toxicity, or withdrawal of consent, whichever happens first.

The maximum duration of BNT314 administration in this study is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to voluntarily give informed consent by signing and dating the informed consent form (ICF) before initiation of any study-specific procedures.
2. Are willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions, and other requirements of the study. This includes that they are able to understand and follow study-related instructions.
3. Are ≥18 years of age at the time of giving informed consent.
4. Have measurable disease according to RECIST v1.1.
5. Have a life expectancy of >3 months.
6. Have Eastern Cooperative Oncology Group Performance Status score of 0 or 1 at screening.
7. Have adequate coagulation function at screening as determined by:

   * International normalized ratio or prothrombin time ≤1.5 × upper limit normal (ULN; unless on therapeutic anticoagulants with values within therapeutic window).
   * Activated partial thromboplastin time ≤1.5 × ULN (unless on therapeutic anticoagulants with values within therapeutic window).
8. Have adequate bone marrow/hematologic function at screening as determined by:

   * Absolute neutrophil count (ANC) ≥1.5 × 10^9/L (≥1500/μL) (patients may not use granulocyte colony stimulating factor or granulocyte-macrophage colony stimulating factor to achieve these ANC levels in the past 7 days).
   * Platelet count ≥100 × 10^9/L (≥100,000/μL).
   * Hemoglobin ≥9 g/dL.
   * Any blood transfusions ≤28 days before first dose of study treatment should be documented.
9. Have adequate hepatic function at screening as determined by:

   * Total bilirubin (Tbili) ≤1.5 × ULN OR direct bilirubin ≤ULN for patients with Tbili levels >1.5 × ULN. Patients with Gilbert's syndrome must have a Tbili <3 mg/dL and direct bilirubin ≤ULN.
   * Alanine aminotransferase and aspartate aminotransferase ≤2.5 ULN for patients with or without liver metastases.
   * Albumin ≥30 g/L.
10. Have adequate renal function at screening as determined by glomerular filtration rate ≥45 mL/min/1.73 m^2 according to the abbreviated Modification of Diet in Renal Disease equation.
11. Have adequate pancreas function at screening as determined by amylase and lipase with no signs and symptoms of pancreatitis.
12. Patients of childbearing potential (POCBP) must have a negative urine or blood beta human chorionic gonadotropin test at screening. Patients that are postmenopausal or permanently sterilized (verified by medical records) will not be considered POCBP, and therefore are not required to undergo pregnancy testing.
13. POCBP must agree to practice a highly effective form of contraception and to require their male partners to use condoms coated with a spermicidal agent, starting at Visit D1 and thereafter until 120 days after receiving the last study treatment.
14. POCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during study, starting at Visit D1 and thereafter until 120 days after receiving the last study treatment.
15. Males who are sexually active and have not had a bilateral vasectomy or orchidectomy must agree to use condoms coated with a spermicidal agent and to require their female partners to practice a highly effective form of contraception during the study, starting at Visit D1 and thereafter until 120 days after receiving the last study treatment.
16. Males must be willing to refrain from sperm donation, starting at Visit D1 and thereafter until 120 days (one sperm cycle) after receiving the last study treatment.
17. Patients must have a histologically confirmed advanced malignant solid tumor, having experienced disease progression on or after standard therapy, or were intolerant of or not eligible for standard therapy.

Other inclusion criteria specific to selected tumor indications may apply.

Exclusion Criteria:

1. Patients that have uncontrolled intercurrent illness, including but not limited to:

   * Ongoing or active infection requiring treatment with anti-infective therapy administered less than 2 weeks prior to first dose.
   * Symptomatic congestive heart failure (Grade III or IV as classified by the New York Heart Association), unstable angina pectoris, or symptomatic untreated cardiac arrhythmia. Treated and/or asymptomatic cardiac arrythmia/atrial fibrillation will be allowed.
   * History of arterial thrombosis or pulmonary embolism within 6 months before the first dose of study treatment.
   * History of myocardial infarction within 6 months before the first dose of study treatment.
   * Uncontrolled hypertension defined as systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg, despite optimal medical management.
   * Prolonged QTc interval at baseline of ≥470 milliseconds using Fridericia's QT correction formula.
   * Ongoing or recent (within one year of screening) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events.
   * History of:

     * Grade 2 immune-mediated myocarditis/colitis/pneumonitis that led to checkpoint inhibitor (CPI) discontinuation. Patients experiencing other Grade 2 immune-mediated adverse events that led to CPI discontinuation, require discussion with the sponsor.
     * Any Grade ≥3 immune-mediated adverse events that led to CPI discontinuation.
     * Patients with Grade 3 adverse events that led to CPI discontinuation but resolved within 21 days without sequalae may also be considered for discussion with the sponsor.
   * History of chronic liver disease (e.g., alcoholic hepatitis or nonalcoholic steatohepatitis, drug-related or autoimmune hepatitis) or evidence of hepatic cirrhosis.
   * History of non-treated intracerebral arteriovenous malformation (shunts), non-treated cerebral aneurysm, spinal cord compression (from disease), carcinomatous meningitis, or stroke will be excluded.
   * History of acute or chronic pancreatitis of any etiology within 6 weeks prior to the start of study treatment.
   * Ongoing pneumonitis or history of noninfectious pneumonitis that has required steroids or evidence of interstitial lung disease.
   * Transient ischemic attack less than one month prior to screening will be excluded.
   * History of brain/central nervous system (CNS) metastases. Patients with newly identified or known unstable or symptomatic CNS metastases will be excluded. Patients with previously treated brain metastases are allowed provided lesions are radiologically stable (i.e., without evidence of progression) for at least 28 days by repeat imaging, latest imaging performed maximum 6 weeks prior to Cycle 1, Day 1.
   * Serious, non-healing wound, skin ulcer (of any grade), or bone fracture will be excluded.
   * Other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation in this clinical study (e.g., acute or chronic pancreatitis, active hepatitis). Known primary immunodeficiencies, either cellular (e.g., DiGeorge syndrome, T-cell negative severe combined immunodeficiency [SCID] or combined T- and B-cell immunodeficiencies (e.g., T- and B-cell negative SCID, Wiskott Aldrich syndrome, ataxia telangiectasia, common variable immunodeficiency).
   * Major surgery within 3 weeks before signature of the ICF unless fully recovered from the surgery in the opinion of the investigator.
   * Any positive test for hepatitis B (defined as positive for hepatitis B surface antigen or hepatitis B virus DNA), indicating acute or chronic infection.
   * Any positive test for hepatitis C (defined as positive for hepatitis C virus antibody or hepatitis C virus RNA), indicating acute or chronic infection.
2. Prior therapy:

   * Radiotherapy within 14 days prior to first BNT314 administration. Palliative radiotherapy will be allowed, but not to target lesions.
   * Any epithelial cell adhesion molecule- or 4-1BB-targeting treatment.
   * Treatment with an anticancer agent within 4 weeks or for systemic therapies after at least five half-lives of the drug, whichever is shorter, prior to study treatment administration.
   * Patient has received any investigational agent (including investigational vaccines) or used an invasive investigational medical device within 28 days before the planned first dose of BNT314 or is currently enrolled in an (another) interventional study. Patients who are in the follow-up phase of an interventional study may participate if they have not received an investigational agent within 28 days (or five half-lives, whichever is longer) of the first dose of BNT314.
   * Patient has a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of the first dose of BNT314. Inhaled or topical steroids, and adrenal or pituitary replacement steroid >10 mg daily prednisone or equivalent, are permitted in the absence of active autoimmune disease.
   * Patient has received granulocyte or granulocyte/macrophage colony stimulating factor (G-CSF/GM-CSF) support within 4 weeks prior to first BNT314 administration or is chronically transfusion dependent; G-CSF and other hematopoietic factors may be used in the management of acute toxicity (such as febrile neutropenia) or prophylactically, when clinically indicated at the investigator's discretion.
   * Received any live vaccine within 30 days prior to the start of study treatment.
3. Known alcohol dependency within 6 months enrollment in this study.
4. Planned enrollment in another study of an IMP, starting after Visit D1 and continuously until the last planned visit in this study.
5. Have a medical, psychological, or social condition which, in the opinion of the investigator, could compromise their wellbeing if they participate in the study, or that could prevent, limit, or confound the protocol specified assessments or procedures, or that could impact adherence to protocol-described requirements.
6. Are subject to exclusion periods from another investigational study.
7. Are vulnerable individuals as per International Council for Harmonisation E6 definition, i.e., are individuals whose willingness to participate in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.
8. Has contraindications (known allergies, hypersensitivity, or intolerance) to the use of BNT314. A patient with a history of hypersensitivity to any component/excipients of BNT314 is also excluded.
9. Are pregnant or breastfeeding and cannot discontinue breastfeeding for the duration of the study and for 4 months after receiving the last dose of BNT314.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity within a cohort | 21 days from the first dose administration
Number and percentage of patients with occurrence of treatment-emergent adverse events (TEAEs) including Grade ≥ 3, serious, fatal TEAE by relationship | from first dose of study treatment to 90 days after last dose of study treatment
  In patients receiving at least one dose of BNT314 per cohort
Number and percentage of patients with occurrence of dose reduction and discontinuation of investigational medicinal product (IMP) due to TEAE | from first dose of study treatment to 90 days after last dose of study treatment
  In patients receiving at least one dose of BNT314 per cohort
Number and percentage of patients with occurrence of Grade ≥ 3 abnormal safety laboratory parameters | from first dose of study treatment to 90 days after last dose of study treatment
  In patients receiving at least one dose of BNT314 per cohort

SECONDARY OUTCOMES:
Geometric means of area under the concentration-time curve from pre-dose to last quantifiable time point prior to the next dose (AUClast) | from pre-dose to 21 days after study treatment for Cycle 1 and Cycle 2
  In patients receiving at least one dose of BNT314 per cohort and are evaluable for PK assessments
Geometric means of area under the concentration-time curve from pre-dose to the end of the dosing period (AUCtau) | from pre-dose to 21 days after study treatment for Cycle 1 and Cycle 2
  In patients receiving at least one dose of BNT314 per cohort and are evaluable for PK assessments
Geometric means of maximum concentration (Cmax) from pre-dose to the end of the dosing period | from pre-dose to 21 days after study treatment for Cycle 1 and Cycle 2
  In patients receiving at least one dose of BNT314 per cohort and are evaluable for PK assessments
Number and percentage of patients who developed detectable anti-drug antibody from baseline to the end of study treatment | from pre-dose to 90 days after last dose of study treatment
  In patients receiving at least one dose of BNT314 per cohort
Disease control rate based on investigator's tumor assessment according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | up to 3 years after first dose of study treatment
  Reported with number and percentage of patients with a confirmed complete response (CR), partial response (PR), or stable disease (SD) (assessed at least 6 weeks after first dose of study treatment) as best overall response. In patients receiving at least one dose of BNT314
Objective response rate based on investigator's tumor assessment according to RECIST v1.1 | up to 3 years after first dose of study treatment
  Reported with number and percentage of patients with a confirmed CR or PR as best overall response. In patients receiving at least one dose of BNT314.
Duration of response (DOR) based on investigator's tumor assessment according to RECIST v1.1 | up to 3 years after first dose of study treatment
  DOR is defined as the time from first objective response (CR or PR) to first occurrence of objective tumor progression or death from any cause, whichever occurs first. In patients receiving at least one dose of BNT314.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (14):
- United States (3):
  - START Midwest, Grand Rapids, Michigan
  - Carolina BioOncology Institute, LLC, Huntersville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
- Belgium (2):
  - GZA Ziekenhuizen, Antwerp
  - CHU de Liège, Liège
- Rigshospitalet, Copenhagen, Denmark
- National Cancer Center Hospital East, Kashiwanoha, Japan
- Spain (4):
  - Hospital Quironsalud Barcelona (NEXT Barcelona), Barcelona
  - Hospital Fund. Jiménez Dia, Madrid
  - Hospital HM Univ. Sanchinarro, Ensayos START, Madrid
  - Clinica Universidad de Navarra, Pamplona
- United Kingdom (3):
  - Royal Marsden Hospital - London, London
  - The Christie Hospital, Manchester
  - Northern Centre for Cancer Care, Newcastle

IPD SHARING:
Plan to Share IPD: No